CLINICAL TRIAL: NCT05858242
Title: Early Auxiliary Diagnosis and Postoperative Recurrence Monitoring of Breast Cancer Based on Plasma ctDNA Methylation Markers
Brief Title: Study on Early Auxiliary Diagnosis and Postoperative Recurrence Monitoring of Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYS-2022002
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: ctDNA methylation; Relapse monitoring
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early and mid-stage breast cancer patients awaiting radical surgery: To explore the predictive effect of plasma ctDNA methylation on postoperative prognosis of breast cancer and the application value of monitoring postoperative recurrence risk through regular postoperative follow-up of stage I-III breast cancer patients undergoing radical surgery.

SUMMARY:
This study screened and identified effective methylation markers in breast cancer, established a detection system for early screening and early diagnosis, and provided a research basis for the embryonic form of non-invasive breast cancer early screening products in later incubation. Then, the plasma ctDNA polygene methylation test was performed for early and middle stage breast cancer patients who were to receive radical surgery for initial treatment, and the predictive effect of postoperative plasma ctDNA methylation status on postoperative prognosis of breast cancer was discussed. In addition, the application value of dynamic monitoring of ctDNA methylation in plasma for postoperative recurrence risk monitoring was explored through regular postoperative follow-up of stage I-III breast cancer patients undergoing radical surgery.

DETAILED DESCRIPTION:
1. This study will be divided into two stages. The first stage will complete the screening, identification, model construction and target verification of polygene methylation markers in the blood of breast cancer patients. The second stage will explore its application in monitoring prognosis and recurrence after radical mastectomy.
2. The first stage (inclusion detection period) : By detecting the DNA methylation characteristics of breast cancer (including tissue and plasma) and non-breast cancer samples (breast tissue/plasma of healthy people, and plasma samples of patients with benign breast lesions), screening, identification and verification of plasma ctDNA polygene methylation markers that can distinguish the differences between breast cancer and non-breast cancer samples are carried out.
3. The second stage (postoperative monitoring and evaluation) : The enrolled group was the initially treated patients who planned to undergo radical mastectomy. Plasma methylation markers were detected before surgery at baseline, and dynamic monitoring of plasma ctDNA polygene methylation detection, related tumor markers and imaging examinations were performed 3 weeks after surgery (or before the start of chemotherapy) and regular follow-up review (once every 3 months for 2 years). To explore the clinical application value of ctDNA methylation status in postoperative breast cancer surgery and follow-up monitoring.

ELIGIBILITY:
The first stage Inclusion Criteria：

Women between the ages of 18 and 80 who are not pregnant or lactating; Meet any of the following categories:

1. Breast cancer Newly diagnosed breast cancer patients [according to breast cancer TNM staging]; The patient was not accepted prior to blood collection Any breast cancer antitumor related treatment, including surgery, transplantation, radiation, chemotherapy, etc.
2. precancerous lesions Dysplasia, carcinoma in situ, atypical hyperplasia, etc., no previous history of malignant tumor.
3. Benign lesions These include fibroadenoma of the breast, intraductal papilloma of the breast, cystic hyperplasia of the breast, lobulated tumors of the breast, Plasma cell mastitis.
4. Healthy people No abnormal breast, no history of malignancy within 5 years; Age 50 years or above.

Exclusion Criteria:

1. previous breast cancer;
2. A history of other cancers;
3. Patients who have received major surgical treatment such as blood transfusion or transplantation within 3 months
4. Participate in other interventional clinical researchers, pregnant or lactating women, or patients suffering from autoimmune diseases, genetic diseases, mental disorders, etc., within 3 months.
5. Patients with other diseases deemed unsuitable for inclusion by the researcher;

The second stage Inclusion Criteria：

1. Patients with definite pathological diagnosis of breast cancer who were to receive radical surgery after preoperative evaluation for initial treatment
2. Women aged between 18 and 80 who are not pregnant or lactating;
3. The radical surgery to be received includes mastectomy radical surgery, simple excision + sentinel lymph node biopsy and modified radical surgery, and on this basis, mastectomy plastic surgery, stage I reconstruction and other operations that have the same radical treatment effect and do not affect the entire standardized treatment of patients
4. Enrolled patients were newly treated breast cancer patients without prior malignant tumor history and treatment history

Exclusion Criteria:

1. Stage IV breast cancer patients, or ECOG score > 2.
2. A history of malignant tumor or other hereditary diseases;
3. Have received organ transplantation, stem cell transplantation, bone marrow transplantation or received blood transfusion within the past month;

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000-1050 samples were used for molecular screening model construction and 100 breast cancer patients awaiting radical surgery were used for 2-year follow-up after treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Finding the characteristic ctDNA methylation targets of breast cancer | assessed up to 36 months
  Establish and verify the early screening model of breast cancer, evaluate the specificity and sensitivity of the model.
To explore the application of postoperative ctDNA methylation in the evaluation of the curative effect of breast cancer surgery and follow-up monitoring | assessed up to 36 months
  The positive and negative prediction rates of ctDNA methylation markers in plasma were analyzed for the recurrence rate 2 years after radical mastectomy for stage I-III breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Rui, Doctor, Principal Investigator — Singlera Genomics Inc.
Locations (1):
- Beijing Friendship Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Oeffinger KC, Fontham ET, Etzioni R, Herzig A, Michaelson JS, Shih YC, Walter LC, Church TR, Flowers CR, LaMonte SJ, Wolf AM, DeSantis C, Lortet-Tieulent J, Andrews K, Manassaram-Baptiste D, Saslow D, Smith RA, Brawley OW, Wender R; American Cancer Society. Breast Cancer Screening for Women at Average Risk: 2015 Guideline Update From the American Cancer Society. JAMA. 2015 Oct 20;314(15):1599-614. doi: 10.1001/jama.2015.12783. PMID 26501536